CLINICAL TRIAL: NCT06832618
Title: A Phase 3b, Double-Blind, Multicenter, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream in Children and Adolescents (6 to <18 Years Old) With Moderate Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of Ruxolitinib Cream in Children and Adolescents (6 to <18 Years Old) With Moderate Atopic Dermatitis
Acronym: TRuE-AD5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB018424-316; 2024-518156-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Ruxolitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Vehicle-controlled (VC) Period: Ruxolitinib (1.5% Cream) (Experimental): Study drug will be administered twice daily.
  Interventions: Drug: Ruxolitinib
- VC Period: Vehicle Cream (Placebo Comparator): Matching vehicle cream will be administered twice daily.
  Interventions: Drug: Vehicle Cream
- Disease Control (DC) Period: Ruxolitinib (1.5% Cream) (Experimental): Study drug will be administered twice weekly.
  Interventions: Drug: Ruxolitinib
- DC Period: Vehicle Cream (Placebo Comparator): Matching vehicle cream will be administered twice weekly.
  Interventions: Drug: Vehicle Cream
- DC Period: Open Label - Ruxolitinib (1.5% Cream) (Experimental): Study drug will be administered twice daily to treat Disease Exacerbations.
  Interventions: Drug: Ruxolitinib
- Open-label Extension (OLE) period: Ruxolitinib (1.5% Cream) (Experimental): Study drug will be administered twice daily.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — The study cream will be applied topically as defined in the protocol for each period.
  Other Names: Opzelura
  Arms: DC Period: Open Label - Ruxolitinib (1.5% Cream); Disease Control (DC) Period: Ruxolitinib (1.5% Cream); Open-label Extension (OLE) period: Ruxolitinib (1.5% Cream); Vehicle-controlled (VC) Period: Ruxolitinib (1.5% Cream)
Drug: Vehicle Cream — Matching vehicle cream will be applied topically as defined in the protocol for each period.
  Other Names: Placebo
  Arms: DC Period: Vehicle Cream; VC Period: Vehicle Cream

SUMMARY:
The purpose of the study is to assess the efficacy and safety of ruxolitinib cream in children and adolescents (6 to <18 Years Old) with moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to < 18 years at the VC Day 1 visit.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria.
* AD duration of at least 3 months for 6 to 11 year olds and at least 2 years for 12 to < 18 year olds (participant/parent/guardian may verbally report signs and symptoms of AD).
* EASI score > 7 at the screening and VC Day 1 visits.
* IGA score of 3 at the screening and VC Day 1 visits.
* Percent BSA (excluding the scalp) with AD involvement of at least 3% and up to 20% at the screening and VC Day 1 visits.
* Itch NRS or WI NRS score ≥ 4 at the screening and VC Day 1 visits, defined as the average of the 7 days directly before the VC/Day 1 visit, with Itch NRS or WI NRS values available for at least 4 of the 7 days.
* Documented recent history (within 12 months before the screening visit) of inadequate response, intolerance, or contraindication to TCSs and TCIs as follows:

  * Inadequate response:

    * For TCSs: Inability of a given TCS to induce and maintain remission or to contain the AD severity at an acceptable level (comparable to an IGA score of 0 [clear] or 1 [almost clear]) despite treatment for 28 days or for the maximum duration recommended by the product prescribing information (eg, 14 days for superpotent TCSs), whichever is shorter and
    * For TCIs: Inability of a given TCI to induce and maintain remission or to contain the AD severity at an acceptable level (comparable to an IGA score of 0 [clear] or 1 [almost clear]) despite treatment according to the product prescribing information.

Note: Documented (within 12 months before the screening visit) systemic treatment for AD (eg, oral corticosteroids, cyclosporine, methotrexate, azathioprine, mycophenolate mofetil) or phototherapy or photo(chemo)therapy can also be considered as a surrogate for inadequate response to TCSs and TCIs.

• Intolerance: Clinically relevant side effects, safety risks, or skin tolerability issues that outweigh the potential treatment benefits and are the reason why a topical treatment could not be restarted or continued.

Note: Documented history (more than 12 months prior to the screening visit) of clinically significant adverse reactions with use of TCSs and/or TCIs that in the opinion of the investigator outweigh the benefits of restarting treatment would also be considered as evidence of intolerance.

• Contraindication: As defined in the product prescribing information.

* Agreement by participants and guardians to discontinue all agents used by the participant to treat AD from the screening visit through the final safety follow-up visit, except as outlined in the protocol.
* For sexually active participants, willingness to take appropriate contraceptive measures to avoid pregnancy or fathering a child for the duration of study participation with the exception of prepubescent participants.

Note: Female participants who have reached menarche must have a negative urine pregnancy test at the screening and baseline visits before the first application of study cream at baseline. They must also take appropriate precautions to avoid pregnancy from the screening visit through the safety follow-up visit.

- Ability to comprehend and willingness to sign an ICF or written informed consent of the parent(s) or legal guardian and a verbal or written assent from the participant when possible.

Note: A signed written ICF must be obtained for inclusion; see protocol.

Exclusion Criteria:

* Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to the VC Day 1 visit.
* Concurrent conditions and history of other diseases as follows:

  * Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome).
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the VC Day 1 visit.
  * Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chickenpox) within 1 week before the VC Day 1 visit.
  * Any other concomitant skin disorder (eg, generalized erythroderma, such as Netherton syndrome), pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
  * Presence of AD lesions only on the hands or feet without prior history of involvement of other classic areas of involvement such as the face or the flexural folds.
  * Other types of eczema within the 6 months prior to screening. Note: Seborrheic dermatitis on the scalp is allowed, as the scalp will not be treated with study cream.
  * Current or history of hepatitis B or C virus infection.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Any of the following clinical laboratory test results at screening:

  * Hemoglobin < 10 g/dL.
  * Liver function tests:

    * Absolute neutrophil count < 1000/μL.
    * Platelet count < 100,000/μL.
    * AST or ALT ≥ 2 × ULN.
    * Alkaline phosphatase > 1.5 × ULN.
    * Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin isfractionated and direct bilirubin < 35%) with the exception of Gilbert disease.
  * Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (using the Modification of Diet in Renal Disease equation).
  * Positive serology test results for HIV antibody.
  * Any other clinically significant laboratory result that, in the opinion of the investigator, poses a significant risk to the participant.
* Use of any of the following treatments within the indicated washout period before the VC Day 1 visit:

  * 5 half-lives or 12 weeks, whichever is longer: biologic agents. For biologic agents with washout periods longer than 12 weeks (eg, rituximab), consult the medical monitor.
  * 4 weeks: systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporine, methotrexate, azathioprine, or other systemic immunosuppressive (eg, JAK inhibitors) or immunomodulating (eg, mycophenolate or tacrolimus) agents.
  * 2 weeks or 5 half-lives, whichever is longer: strong systemic CYP3A4 inhibitors.
  * 2 weeks: immunizations with live-attenuated vaccines; sedating antihistamines unless on a long-term stable regimen (nonsedating antihistamines are permitted).

Note: COVID-19 vaccination is allowed.

• 1 week: use of other topical treatments for AD, other than bland emollients (eg, Aveeno® creams, ointments, sprays, soap substitutes), such as antipruritics (eg, doxepin cream), corticosteroids, calcineurin inhibitors, PDE4 inhibitors, coal tar (shampoo), antibiotics, or antibacterial cleansing body wash/soap.

Note: Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week and their frequency remains the same throughout the study.

* History of treatment failure with any systemic or topical JAK inhibitor (eg, ruxolitinib, tofacitinib, baricitinib, abrocitinib, upadacitinib) for AD or any other inflammatory condition.
* Ultraviolet light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 2 weeks prior to the baseline visit and/or intention to have such exposure during the study that is thought by the investigator to potentially impact the participant's AD.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before baseline with another investigational medication or current enrollment in another investigational drug Protocol.
* Pregnant or lactating participants or those considering pregnancy during the period of their study participation.
* Living with anyone participating in any current Incyte-sponsored ruxolitinib cream study.
* Known allergy or reaction to any component of the study cream formulation.
* In the opinion of the investigator, unable or unlikely to comply with the administration schedule, study evaluations, and procedures (eg, eDiary compliance).
* Committed to a mental health institution by virtue of an order issued either by the judicial or the administrative authorities.
* Employees of the sponsor, sponsor delegates (eg, contract research organizations), or investigators or are otherwise dependents of them.
* The following participants are excluded in France: vulnerable populations according to article L.1121-6 of the French Public Health Code and adults under legal protection, or who are unable to express their consent per article L.1121-8 of the French Public Health Code, not affiliated to a social security per article L.1121-8-1 of the French Public Health Code.
* In the EU, participants considered incapacitated (according to CTR Article 31).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2028-05-18 (Estimated)

PRIMARY OUTCOMES:
VC Period: Binary response status of Eczema Area and Severity Index 75 (EASI75) | VC Week 8
  Defined as achieving ≥ 75% improvement in Eczema Area and Severity Index (EASI) score from baseline.

SECONDARY OUTCOMES:
VC Period: Binary response status of Investigator's Global Assessment Treatment Success (IGA-TS) | VC Week 8
  Defined as achieving Investigator's Global Assessment (IGA) score of 0 or 1 with ≥ 2-grade improvement from baseline.
VC Period: Binary response status of ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | VC Week 8
  Defined as achieving ≥ 4-point improvement in Itch NRS [participants aged 12 to < 18 years] or Worst Itch Numerical Rating Scale (WI NRS) [participants aged 6 to < 12 years] score from baseline.
DC Period: Time to first disease exacerbation, defined as Investigator's Global Assessment score of ≥ 2 (DE) in the DC period | Up to 44 Weeks
  Defined as responders [IGA score < 2] from the VC period or the OLE period rerandomized to proactive treatment, time to first DE, where DE is defined as IGA score of ≥ 2.)
Number of Treatment Emergent Adverse Events (TEAEs) | From Baseline up to 70 weeks
  Defined as any AE reported for the first time or worsening of a pre-existing event after the first application of study cream.
Binary response status of Eczema Area and Severity Index 75 (EASI75) at each postbaseline visit except Week 8 | Up to 44 weeks
  Defined as achieving ≥ 75% improvement in Eczema Area and Severity Index (EASI) score from baseline.
Binary response status of Investigator's Global Assessment Treatment Success (IGA-TS) at each postbaeline visit except Week 8 | Up to 44 weeks
  Defined as achieving Investigator's Global Assessment (IGA) score of 0 or 1 with ≥ 2-grade improvement from baseline.
Binary response status of ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Days 2, 3, and 7 and VC Weeks 2 and 4
  Defined as achieving ≥ 4-point improvement in Itch NRS [participants aged 12 to < 18 years] or Worst Itch Numerical Rating Scale (WI NRS) [participants aged 6 to < 12 years] score from baseline.
VC Period: Time to achieve ITCH4 | Up to 8 weeks
  Defined as time to achieve ≥ 4-point improvement in Itch NRS [participants aged 12 to < 18 years] or Worst Itch Numerical Rating Scale (WI NRS) [participants aged 6 to < 12 years] score from baseline.
VC Period: Binary response status of both EASI75 and IGA-TS at each postbaseline visit in the VC period | Up to 44 weeks
VC Period: The binary response status of DLQI-4/CDLQI-4 at VC Weeks 2, 4, and 8 | Weeks 2, 4 and 8
  Dermatology Life Quality Index (DLQI)-4/ Children's Dermatology Life Quality Index (CDLQI)-4 is defined as achieving ≥ 4-point improvement in DLQI/CDLQI from baseline.
VC Period and DC Period: Change from baseline in the CDLQI (or DLQI) score at each postbaseline visit | Up to 52 weeks
  The DLQI will be administered to participants aged 16 and 17 years. The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. The CDLQI will be administered to participants aged 6 to 15 years. The CDLQI is a simple validated questionnaire to measure how much the skin problem has affected the participant over the past week (7-day recall). The higher the score, the more quality of life is impaired.
VC Period and DC Period: Change from baseline in the Patient-Oriented Eczema Measure (POEM) score at each postbaseline visit | Up to 52 weeks
  The POEM is a 7-question quality-of-life assessment that asks how many days the participant has been bothered by various aspects of their skin condition during the past 7 days. A negative change from Baseline indicates improvement.
VC Period and DC Period: Acceptability and tolerability assessment (exit interview/questionnaire) | VC Period Week 8 and DC Period Week 44
  The overall impression of the acceptability and tolerability of study cream will be assessed quantitatively using the Pediatric Impression of Cream Acceptability and Tolerability questionnaire. This is a structured questionnaire with 2 questions: one for assessing overall impression of acceptability and one for assessing tolerability. Each question has 4 possible response options, with a corresponding score from 1 to 4. The total score will range from 2 (most acceptable and tolerable) to 8 (least acceptable and tolerable).
DC Period: Number of disease exacerbations (DEs) | Up to 44 weeks
  Defined as Investigator's Global Assessment score of ≥ 2.
DC Period: Amount of ruxolitinib cream used | Up to 44 weeks
VC Period: Plasma concentrations of ruxolitinib and PK parameters (Ctrough,ss) | VC Week 2 and VC Week 8
  Trough and steady-state concentrations for ruxolitinib in plasma will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (96):
- United States (20):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Saguaro Dermatology, Phoenix, Arizona
  - National Jewish Health, Denver, Colorado
  - Encore Medical Research, Llc Hollywood, Hollywood, Florida
  - Lane Dermatology and Dermatologic Surgery, Columbus, Georgia
  - Cleaver Medical Group, Cumming, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Sneeze Wheeze and Itch Associates Llc, Normal, Illinois
  - Endeavor Health Medical Group, Skokie, Illinois
  - Raven Clinical Research, Marriottsville, Maryland
  - Oakland Hills Dermatology Pc, Auburn Hills, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Red River Research Partners, Bolivar, Missouri
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University of Texas Physicians - Bellaire Station, Bellaire, Texas
  - Frontier Dermatology, Mill Creek, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (6):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Az Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Grand Hôpital de Charleroi-Les Viviers, Gilly
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Dermatologie Maldegem, Maldegem
- Canada (14):
  - Kirk Barber Research, Calgary, Alberta
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Laster Rejuvenation Clinics Edmonton D.T. Inc., Edmonton, Alberta
  - Dr. Chih-Ho Hong Medical Inc., Surrey, British Columbia
  - University of British Columbia (Ubc) - British Columbia Children'S Hospital (Bc Children'S Hospital), Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Leader Research, Hamilton, Ontario
  - Facet Dermatology, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Centre de Recherche Saint-Louis, Montreal, Quebec
  - Chu Sainte-Justine, Montreal, Quebec
  - Chu de Quebec Universite Laval, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
  - Skincare Studio Dermatology Centre, St. John's
- France (3):
  - Bordeaux Chu Hopital Saint - Andre, Bordeaux
  - Polyclinique Reims-Bezannes, Reims
  - Hopitaux Drome Nord, Romans-sur-Isère
- Germany (9):
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim
  - Universitatsklinikum Bonn Aoer, Bonn
  - Drk Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - Universitaetsklinikum Carl Gustav Carus Tu Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatsmedizin Goettingen, Göttingen
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitatsklinikum Munster, Münster
- Hungary (8):
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Geomedical Orvosi Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpon Belgyogy Klinika, Debrecen
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Aok Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Italy (5):
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico San Marco, Catania
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Azienda Ospedaliera Universitaria Federico Ii, Naples
  - Azienda Ospedale Universita Di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Rome
- Umc Utrecht, Utrecht, Netherlands
- Poland (14):
  - Centrum Badan Klinicznych Pi-House Sp. Z O.O., Gdansk
  - Gyncentrum Sp. Z O.O., Katowice
  - Grazyna Pulka Centrum Medyczne All Med Spolka Komandytowa, Krakow
  - Diamond Clinic Sp. Z O.O., Krakow
  - Dermoklinika, Lodz
  - Clinical Best Solutions Sp. Z O.O. Sp. K., Lublin
  - Dermodent Centrum Medyczne Czajkowscy S.C., Osielsko
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Mics Centrum Medyczne Toruń, Torun
  - Mics Centrum Medyczne Warszawa Chlodna, Warsaw
  - High-Med Przychodnia Specjalistycza, Warsaw
  - Centrum Medyczne Evimed, Warsaw
  - Etg Warszawa, Warsaw
  - Dermmedica Sp. Z O.O., Wroclaw
- Spain (10):
  - Hospital General Unviersitario de Alicante, Alicante
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital de Manis, Manises
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
- United Kingdom (6):
  - West Glasgow Ambulatory Care Hospital, Glasgow
  - St John'S Institute of Dermatology, London
  - The Adam Practice, Metropolitan Borough of Wirral
  - University of Nottingham Health Service, Nottingham
  - Sheffield Childrens Hospital, Sheffield
  - Walsall Manor Hospital, Walsall

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to assess the efficacy and safety of ruxolitinib cream in children and adolescents (6 to <18 Years Old) with moderate atopic dermatitis — https://incyteclinicaltrials.com/studies/incb018424-316